# ClinicalTrials.gov

de Mama Estadios I-III.

**Protocol Registration and Results System (PRS)** ClinicalTrials.gov ID: [Not yet assigned] Last review date: October 13th, 2023. Study Identification Unique Protocol ID: 023-005-OMI(CEI-05022) Brief Title: Improving Lifestyle Behavior by "Joven, Fuerte y Saludable" Multidisciplinary Program. Official Title: Efecto de Una intervención Multidisciplinaria de Estilo de Vida Sobre el Exposoma de Pacientes premenopáusicas Con cáncer 

- 16 **Title:** Improving Lifestyle Behavior by "Joven, Fuerte y Saludable" Multidisciplinary
- 17 Program. Official Title: Efecto de Una intervención Multidisciplinaria de Estilo de Vida
- Sobre el Exposoma de Pacientes premenopáusicas Con cáncer de Mama Estadios
- 19 I-III.

20

# <u>Abstract</u>

- Background. Breast cancer (BC) is the leading cause of cancer-related death and 21 22 disability in young women. Patients with BC experience physical symptoms and psychosocial distress that adversely affect their quality of life (QoL), physical 23 functioning, and psychological well-being. "Joven & Fuerte" is a navigation program 24 for young women with BC at the National Cancer Institute in Mexico City. The 25 program proposes an hybrid model (face-to-face and virtual) to support patients on 26 aspects such as oncology, nutrition literacy, and psychology with mindfulness. 27 **Methods.** The study was initially planned as a randomized controlled trial to ensure 28 accurate results. However, during the pilot study, it was adapted to meet the specific 29 30 needs of patients such as oncology consultations and in consideration of living arrangements. Two groups will be compared: one receives hybrid education and the 31 other, a hybrid education and personalized intervention. Patients who agreed for the 32 face-to-face sessions were assigned to the personalized interventions group, and 33 34 others, to the hybrid education group. The intervention group receives an in-person consultation to evaluate their physical measurements and an interdisciplinary 35 assessment by experts. Patients can ask for virtual assistance through Zoom and 36 WhatsApp in case of any issues during the intervention. In addition, educational 37 materials such as healthy lifestyle guides and videos can be accessed through 38 39 Facebook and YouTube groups upon request. To ensure the comprehension of the material, follow-up sessions are conducted through phone calls, video calls, or on-40 site visits. Validated questionnaires will assess lifestyle habits, QoL status, and 41 42 levels of distress, anxiety, and depression.
- What is already known on this topic
  - Breast cancer and its treatment impacts the lifestyle and quality of life of patients.
    - Improvement in nutrition, lifestyle, and psychological wellbeing positively impacts the prognosis of breast cancer and quality of life or survivors.
- 48 What this study adds

44

45

46

47

49

50

- Provides interventions for patients living far from a hospital.
- Evaluates the health advantages of educational and personalized interventions.

- Examines how lifestyle changes affect the quality of life, mental health, and physical functioning of patients with breast cancer receiving cancer treatment.
- How this study might affect research, practice, or policy
  - This hybrid approach is both viable and economical for public institutions.
    - The findings of this study will reveal the effects of these interventions and their potential benefits to patients.

#### INTRODUCTION

52 53

55

56

57

- Breast cancer (BC) is a leading cause of death in women worldwide, especially in 59 Latin America, where patients often present with advanced stages of aggressive 60 61 subtypes of BC at a younger age (1). The risk of BC depends on various factors, 62 including hormone replacement therapy history, reproductive history, alcohol or tobacco consumption, physical activity, and dietary habits, that are collectively called 63 exposome (2). Exposome refers to the exposure to environmental influences and 64 biological responses throughout a person's life from the prenatal stage. It can be 65 66 influenced by the environment, diet, behavior, and endogenous processes (3).
- External exposome refers to environmental factors such as mental stress, climate, 67 and lifestyle. In contrast, internal exposome are changes within an organism such 68 as increased stress hormones, inflammatory cytokines, and oxidative stress (4). 69 70 Constant exposure to environmental factors, such as an unhealthy lifestyle, can cause cellular damage and contribute to the growth and evolution of tumors. Once 71 72 cellular damage occurs, internal exposome promotes changes that create a harmful environment, favoring cancer cells to acquire mechanisms to cope with stress and 73 drugs, leading to a resistance to oncological treatments (5). 74
- Obesity is part of the personal exposome and can impact the internal exposome, 75 potentially affecting BC patients. A significant percentage of patients diagnosed with 76 BC (70.9%) are overweight or obese at the time of diagnosis (6). This weight gain 77 78 usually occurs during systemic treatment, with 25% of patients gaining weight within six months, 32% between 6-12 months, and 20% between 12-18 months after 79 diagnosis (7). Young women with breast cancer (YWBC) also experience and 80 increase in weight since the initiation of oncological treatment and up to the second 81 82 year of diagnosis (from 39% at baseline to 46% in two years), highlighting the importance of evaluating the implications of weight gain and whether early 83 intervention would help control the risk factors mentioned earlier (8). Obesity may 84 also be associated with worse disease-free and overall survival (9). 85

Weight gain in patients with BC is often associated with several factors, including systemic treatment, diagnosis at a young age, and lifestyle changes resulting from the disease or treatment. However, the primary mechanism underlying weight gain is reduced physical activity (10). The combination of chemotherapy and endocrine therapy is linked to higher weight gain, especially in patients who are premenopausal (a gain of up to 24 kg). In contrast, those who are postmenopausal tend to lose weight (11).

BC patients have reported experiencing physical symptoms and psychological 93 distress, which can negatively impact their quality of life (QoL). These symptoms can 94 95 affect their physical functioning, psychological well-being, and social support levels (12). Particularly, YWBC is a vulnerable population with specific concerns such as 96 fertility, self-image, QoL, sexuality, and personal goals (13) and experience high 97 anxiety and depression (14). Maintaining a healthy lifestyle can improve QoL and 98 99 lead to better prognoses and lower mortality rates (15). For example, exercise can reduce breast cancer-related death risk by 30% and all-cause death risk by 41% 100 (16). Patients undergoing oncology treatment face various nutritional challenges that 101 differ based on the type and stage of cancer, and the treatments may worsen these 102 challenges. Early nutritional screening and interventions are crucial in the cancer 103 104 population, as emphasized in the clinical guidelines (ASPEN/ESPEN) (17).

The Instituto Nacional de Cancerología (INCAN) in Mexico City offers a program 105 called "Joven & Fuerte" for young women diagnosed with BC. However, the attention 106 107 was not systematic and it was difficult to measure the benefits of the intervention. So the present study proposes a psychological intervention, side effect management, 108 109 physical activity, sleep hygiene, and psychological strategies, with onsite and remote interventions to improve patient adherence and ensure timely attention. The study 110 111 aims to evaluate the impact of early intervention on metabolic control in newly diagnosed BC patients, their QoL, and clinical outcomes. 112

#### **METHODS**

- A controlled trial design was adopted in which patients were assigned to two intervention groups according to the nutritional, psychological, or rehabilitation risk at baseline or according to their geographical localization. The first group will receive a hybrid multidisciplinary lifestyle education intervention, whereas the second group will receive an individualized hybrid multidisciplinary lifestyle intervention.
- For sample size estimation, we used internal statistics from the Mammary Tumor Department at the INCAN, which has an annual average of 109 women diagnosed and treated based on the selection criteria. Considering the effect on metabolic and inflammatory parameters, a study by Dieli-Conwright et al. (18) was followed to

- identify the difference in the decrease in insulin parameters by 14%. A confidence
- level of 95% and power of 80% were considered with a control: intervention ratio of
- 1:1. Thus, a sample size of 132 patients was obtained. Considering a probable loss
- of 10%, 146 patients were invited to participate in the study, with 73 patients per
- 127 group.

128

133

134

135

136

137

138

139140

141

142

143

144

145

146147

148

149

151

156

#### Inclusion criteria

- Women aged ≥18 and <40 years who were diagnosed with stage I-III BC,</li>
   confirmed by pathology and image at the INCAN
- Candidates for multidisciplinary treatment, including surgery, chemotherapy, and/or hormonal treatments.
  - Signed the informed consent form
  - Have access to a mobile phone or any electronic device with an active internet connection to receive the program information.

#### **Exclusion criteria**

- Patients with inflammatory cancer
- Those with cardiomyopathy or ventricular dysfunction (NYHA >II), arrhythmia secondary to left ventricular ejection alterations that require medication, previous myocardial infarction, or angina pectoris in the last six months
  - Receiving treatment for cardiovascular or cerebrovascular disease, inflammatory bowel disease, malabsorption syndrome, rheumatoid arthritis, lupus, thyroid diseases, or Cushing syndrome
  - Unable to walk for at least 1 km
  - Have cardiovascular, respiratory, or musculoskeletal diseases that impede physical activity
  - Pregnant or breastfeeding
- Have psychiatric conditions impeding active participation in this protocol
- Do not understand Spanish

#### Selection and group assignment of the patients

- Patients will be recruited through an active program at the INCAN, where potential
- candidates will be identified and invited by the navigator at the program "Joven &
- Fuerte." After they sign the informed consent form (ICF), patients will be assigned
- into one of the two groups:
  - Group 1: Hybrid multidisciplinary lifestyle education intervention.

# Group 2: Individualized hybrid multidisciplinary lifestyle interventions.

The initial proposal was randomized assignment to each group; however, the pilot study revealed challenges for patients who lived far from the hospital, in other states, or had personal obligations such as family or work. Therefore, the randomization process was adapted to meet the patients' needs. The intervention aims to facilitate patients' adherence and follow-up with healthcare providers. Additionally, patient preferences were considered when assigning them to a group.

#### Intervention

157

164

177

178

179

180 181

182

183

184 185

186

The individualized hybrid multidisciplinary lifestyle intervention consists of four 165 phases. During the initial phase, (1st month), patients undergo psychological, 166 nutritional, and physical evaluations using validated questionnaires. Weekly follow-167 168 ups are scheduled to answer any questions and provide educational materials. Psychological intervention for the management of stress, anxiety, or other sleep 169 disorders begins during this phase. Changes in diet and physical activity levels are 170 prepared based on baseline questionnaires and adjusted to their needs and 171 preferences to facilitate adherence to the intervention. Basic nutritional orientation is 172 provided covering topics such as identification of food groups using guides such as 173 "My Plate" (19) from the American Association of Diabetes, how to read nutrition 174 facts labels, and explanation on following a healthy diet, with available food groups 175 in the country. 176

In the **consolidation phase**, from second to sixth month, patients undergo follow-ups every two weeks on-site or remotely, depending on the patient's preference. Follow-up was to monitor patients' symptoms and adjust their diet and exercise routines accordingly. Psychological intervention will be tailored to individual needs if a patient experiences symptoms such as nausea, vomiting, diarrhea, or fatigue. This phase aims to help patients become independent and manage their activities without professional help. A personalized diet and exercise plan will be created for each patient, considering their socioeconomic status. The local food groups available to each patient are prescribed. The Avena Health application will monitor water consumption, physical activity, and nutritional adherence if the patient has access.

The **maintenance phase**, from seventh to 12<sup>th</sup> month, the patients will be followed up every two months. Anthropometric measures, blood tests, and questionnaires will be used to assess their progress. The objective of this phase is to reinforce the recommendations of previous phases.

The patients undergo check-ins every three months during the follow-up phase, which begins after 12 months. In the medium term, anthropometric measures and

questionnaires will be used to evaluate patient adherence to multidisciplinary interventions. Any questions or concerns will be addressed during the checks. See **Figure 1.** 



Created in **BioRender.com** bio

Figure 1. Joven, Fuerte y Saludable, Protocol Design.

# Components of the Multidisciplinary Individualized Intervention

#### 199 Nutritional Intervention

Patients will undergo a comprehensive nutritional assessment and receive guidance on maintaining a healthy diet balanced with macronutrients. Assessment of symptoms that affect nutritional or metabolic status; anthropometric indicators such as weight, height, waist circumference, arm circumference, waist-to-hip ratio, and body composition determined by bioelectrical impedance analysis (BIA) will be collected at baseline and follow-up; and biochemical parameters such as blood glucose, insulin, HbA1c, total, low-density lipoprotein-cholesterol, high-density lipoprotein-cholesterol, triglycerides, and c-reactive protein (CRP) will be assessed. Recommendations will be tailored to the individual's needs and budget and any adverse effects related to their cancer treatment, focusing on a healthy, moderately hypocaloric diet (for those who are overweight, obese, or at metabolic risk) or an isocaloric diet for those who are underweight, considering the individualized requirements of energy, protein, carbohydrate, lipids, vitamins, and minerals. Dietetic assessment measures adherence to the diet prescription through a typical

- 214 feeding model or 24-hour recall. Participants will meet the program nutritionist
- 215 according to the visit frequency described for each phase.
- A webpage will be available with weekly modules on nutrition, and patients will be
- invited to workshops to resolve any obstacles they encounter while implementing
- 218 recommendations. A virtual class would be offered if someone could not attend the
- workshop. A workbook with educational information and a diary section will also be
- 220 provided, allowing patients to share their thoughts on the intervention, challenges
- they face, and questions.
- 222 Physical activity intervention
- 223 Patients will be prescribed a customized regimen of dynamic aerobic exercise to
- improve their physical capacity. A stress test determines maximum effort capacity
- 225 and identifies contraindications. The rehabilitation team will evaluate the
- 226 performance status of patients using the Karnofsky Index (a functional scale) and
- 227 Eastern Cooperative Oncology Group (ECOG). Patients receive personalized
- treatment based on their diagnoses. In addition, they will receive a digital or physical
- 229 guide of exercises appropriate for their disease stage. They should perform these
- exercises 3-5 times weekly for at least 150 minutes, including resistance training and
- 231 moderate-intensity aerobics. Patients with special needs, such as those with
- lymphedema, post-surgery, or active treatment, can also undergo various exercises.
- A healthcare professional trained in oncological rehabilitation will supervise all the
- 234 exercise sessions.
- 235 Psychological intervention
- During the diagnosis and treatment of BC, workshops will be held in collaboration
- with a psychology team to assess the emotional symptoms. Patients will receive
- videos of relaxation techniques and their anxiety levels will be monitored using a
- thermometer anxiety tool. Patients who score more than four will complete
- depressive and anxiety symptom questionnaires (the Patient Health Questionnaire,
- 241 PHQ-9 and Generalized Anxiety Disorder, GAD-7, respectively) and will be referred
- for group or individual therapy. The number of therapy sessions will be limited to
- 243 eight for individual interventions and two for each multidisciplinary intervention
- 244 phase. The questionnaires will be administered at the beginning and at three, six,
- 245 nine, and 12 months.
- 246 Psychological interventions will involve cognitive-behavioral therapy, which will focus
- on changing cognition and behaviors to reduce symptoms of stress, anxiety, and
- 248 depression. Treatment will also address the emotional discomfort caused by the
- 249 diagnosis and treatment and its impact on family and couple dynamics, social and

250 work life, body image, sexuality, and fertility etc. During the sessions, a clinical history will be taken, with which a Clinical Map of Pathogenesis and Goal Scope Map 251 252 will be generated according to the Nezú and Nezú model (4). This assessment 253 allows the development of a therapy focused on the patient's needs and, to identify 254 intervention strategies for achieving specific goals, such as psychoeducation, relaxation training, cognitive restructuring, problem-solving therapy, behavioral 255 activation, and assertive communication training. Patients can choose between 256 hybrid formats such as Zoom and WhatsApp and onsite sessions with specialists. 257

#### 258 Mindfulness + oncologic rehabilitation intervention

The oncological rehabilitation and mindfulness program consists of four modalities:

- Group face-to-face,
- Individuals face-to-face
- Group online, and
- Individual online

259

272

- The program can be applied at different time points during patient treatment: before, after, and after surgery with chemotherapy and/or radiotherapy.
- Physical exercises include different activity levels for patients to improve their flexibility, range of motion, strength, and recovery capacity; exercises included in the program are aimed at working different parts of the body, combined into different techniques divided into static, moving, breathing, and meditation techniques, and Thai-Chi and Qi Gong, as part of the mindfulness program. The contents of the program are presented in **Table 1**.

# Table 1. Mindfulness and oncologic rehabilitation content

| PROGRAM<br>ADMISSION | ONCOLOGIC<br>REHABILITATION | EXERCISES | MOVEMENT<br>TECHNIQUES | STATIC<br>TECHNIQUES | BREATHING<br>TECHNIQUES | MEDITATION<br>TECHNIQUES | EDUCATIONAL<br>MATERIAL |
|---|---|---|---|---|---|---|---|
| Interview (E) | Flexibility (RFi) | Neck (C) | Expansion and contraction (ECS) | Body scan (on<br>the floor) (EA) | Conscious<br>breathing<br>(RCS) | Static<br>meditation<br>(ME) | Welcome to the program! (BVP) |
| Initial<br>evaluation<br>(EI) | Range of movement (RRM.ii) | Upper limbs (MS) | Expansion<br>and<br>contraction on<br>the wall (ECP) | Body scan<br>(seated) <b>(ES)</b> | Conscious<br>breathing (5<br>words)<br>(RCS5) | Static<br>meditation<br>(seated)<br>(MES) | Benefits of oncologic rehabilitation (BFRO) |

| Questionnaire<br>application<br>(AC) | Strength (Rfza. III) | Lower limbs (MI) | 21 movements (21M) | Internal<br>circulation<br>channel (CIC) | Breathing<br>awareness<br>(chest, costal,<br>abdominal)<br>(RAWS) | Lay down<br>meditation<br>(MA) | Benefits of<br>mindfulness<br>(BFAP) |
|---|---|---|---|---|---|---|---|
| Postural<br>hygiene ( <b>HP</b> ) | Recovery (RR.IV) | Legs (P) | Tai Chi's 13<br>movements<br>(13M) | | Abdominal breathing (RA) | Walking<br>meditation<br>(MC) | Stress<br>consequences<br>(CSCE) |
| Integration of<br>the program<br>(IP) | | Thorax (T) | 5 animals (Qi<br>Gong) <b>(5A)</b> | | Breath count (CR) | Moving<br>meditation<br>(MCM) | Cortisol (CZ) |
| Psychological intervention (IPS) | | Hip <b>(H)</b> | | | | | Sixth sense (SS) |
| | | | | | | | Nutrition (NT) |

273 \*Codes used in this intervention are marked in bold and in parentheses.

- 275 Finally, sessions will be completed by ensuring that the patients are aware of the
- importance of how stress impacts health, reminding them that specific at-home
- exercise techniques could improve their physical condition.
- 278 Educative intervention
- 279 Psychologic and mindfulness educative intervention
- Virtual educational intervention was adjusted to STREAM intervention for BC after
- 281 adapting it for our population (20). Based on our experience with the Joven & Fuerte
- program this intervention with continue for 10 weeks, from the beginning of the
- diagnosis, which, is when the patient requires understanding and assimilating their
- 284 diagnosis and the life changes that cancer treatments will represent, as well as adapt
- to the institution. This intervention intends to manage the emotional stress of this
- 286 phase in collaboration with the psychology and mindfulness team.
- Questionnaires will be administered to evaluate QoL (QLQ-C30 and QLQ-BR23) at
- 288 the baseline and at three, six, 12, and 18 months, and healthy lifestyle (WCFR/AICR)
- at the beginning and end of the intervention in both groups.

While these activities are performed, patients will participate in a mindfulness workshop for 10 weeks, which includes breathing counting techniques (Zazen), guided meditations (five words of self-composure), meditation exercises with static movement (BaDuanJin), conscious walking (Kinjun), body scan, energy concentration work and physical movement (five healing animals), moving meditation (TaiChi), and yoga. All of these techniques are intended to be tools for the patient to deal with the stress she faces during her BC diagnosis.

# Healthy lifestyle educative intervention

The healthy lifestyle education intervention was adapted from the Diabetes Prevention Program (DPP)(21) funded by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) and has been used in BC studies, such as SUCCESS (22), MEDEA (23), and PASAPAS (24). This educational material is planned to be given to all intervention groups. Every week, in a hybrid format, patients will receive a WhatsApp or, through the Facebook group, the written information, video, and/or audio of the subjects included in the program. Additionally, patients will receive a manual with a weekly description of the topic to be discussed and the activities they must carry out that week in a way that the patient will have the whole week to carry out her activities; on Friday, a session will be opened both on Zoom or WhatsApp, or in the case of patients who can physically go to the institute in person. The expert will also be available so that the patient can share her doubts and difficulties faced during the week.

On **Table 2**, educational subjects reviewed on every intervention phase are described.

| Intervention phase | Follow-up | Week | Title | Content |
|---|---|---|---|---|
| Intensive phase: weekly follow-up | 1 | 1 | Welcome to the program | Introduction |
| | 2 | 2 | Caloric balance | Caloric restriction |
| | 3 | 3 | Type of fatty acids | Caloric restriction |
| | 4 | 4 | Reducing calories, controlling portions | Caloric restriction |

| | 5 | 5 | Muscular movement | Physical activity |
|---|---|---|---|---|
| | 6 | 6 | Working with your surroundings | Behavioral support |
| | 7 | 7 | Problem-solving | Behavioral support |
| | 8 | 8 | Being active: a way of living Physical activ | |
| | 9 | 9 | Healthy eating | Caloric restriction |
| | 10 | 10 | Healthy eating and breast cancer | Breast cancer and nutrition |
| | 11 | 11 | Preparing a better breakfast, Caloric restriction lunch, and dinner behavioral support | |
| | 12 | 12 | Progress review | Recap and evaluation |
| Consolidation phase:<br>two-week follow-up | 13 | 14 | Answering negative thoughts | Behavioral support |
| | 14 | 16 | The slope in changing to a healthy lifestyle | Behavioral support |
| | 15 | 18 | Intensifying physical activity | Physical activity |
| | 16 | 20 | 10 ways to control hunger | Behavioral support |
| | 17 | 22 | What to eat on holidays | Behavioral support |
| | 18 | 24 | Making balance and celebrating success | Recap and evaluation |
| | 19 | 28 | How to stay motivated | Behavioral support |

| Maintenance phase:<br>monthly follow-up | 20 | 32 | Recovering from excess eating | Behavioral support |
|---|---|---|---|---|
| | 21 | 36 | Weight loss review | Caloric restriction |
| | 22 | 40 | How to adapt to long-lasting success | Behavioral support |
| | 23 | 44 | Preparing for what's yet to come | Recap and evaluation |
| | 24 | 48 | Congratulations! You finished the program! | Recap and evaluation |

# Table 2. Intervention phases adapted from the diabetes education program (DPP)

# Barriers and facilitators for the multidisciplinary program implementation

As this program is being implemented for the first time and with the aim of enhancing patient care, the assessment of barriers will be carried out through questionnaires administered to both program staff and enrolled patients. The purpose is to identify the barriers faced by each party, thereby enabling the provision of solutions alongside the interventions. The questionnaire design was based on the CFIR/RE-AIM framework, a tool used to assess the success of program implementation (25, 26).

# Data analysis

314

315

323

332

333

334

335

Descriptive statistics will be performed for the clinical and demographic data. 324 Inferential comparisons will be made by calculating the relative risk with 95% 325 326 confidence intervals. To compare the effect between groups, a statistical comparison with the Kolmogorov-Smirnov test will be performed, and depending on the 327 distribution of data, parametric (normal distribution) or non-parametric (non-normal 328 distribution) tests will be applied. To evaluate the differences between groups, 329 330 Student's T test for related groups or the Mann-Whitney test will be used, while for the analysis of repeated samples, analysis of variance (ANOVA) will be used for 331

three or more variables, depending on the nature of the data.

Chi-square and Fisher's tests will be used to compare categorical variables, and the alpha value will be set to 0.05. Bivariate analysis will be performed to identify differences between groups and associations with survival concerning the measured

clinical variables and biomarkers. To analyze the existing correlation with the clinical variables, Pearson or Spearman regression with a 95% confidence interval will be used, depending on the nature of the data distribution. To determine the associations between independent variables, multivariate logistic regression models were used, adjusting for the remaining clinical variables.

#### Discussion

Although various interventions provide nutritional and physical activity counseling, most of them are focused on patients who have survived cancer and do not include those who have been diagnosed recently. Emotional support is also not taken into account. A recent meta-analysis published by Cochrane reviewed 20 studies and involved 2028 patients with breast cancer who received interventions for weight loss. The results showed that these interventions for survivors of breast cancer with obesity resulted in moderate weight reduction, improved body mass index and waist circumference, and enhanced quality of life through diet and exercise interventions (7). It appears that a multidisciplinary approach could lead to even better results, and probably it has to be since the diagnosis to start a mentality switch since the beginning of the disease.

Nutritional interventions in patients with cancer ensure adequate intake of energy and nutrients during oncological treatment, which results in an improved response and reduced toxicity of pharmacological anti-cancer therapies. These health changes reduce the long-term side effects of treatment and promote long-term overall health (27). The Women's Intervention Nutrition Study (WINS) demonstrated the impact of nutritional intervention on the prognosis and survival of BC, with a low-fat diet promoting modest weight loss, improving metabolic biomarkers, and positively affecting disease-free survival (28). According to lifestyle guidelines recommended by the World Cancer Research Fund (WCRF)/American Institute for Cancer Research (AICR), a fiber- and soy-rich diet and limited consumption of fatty acids (especially saturated fatty acids) can improve survival after BC diagnosis (27).

According to research by Demark-Wahnefried et al., women undergoing chemotherapy may experience a decrease in energy expenditure due to reduced activity despite same calorie intake (29). The Health, Eating, Activity, and Lifestyle (HEAL) study also found that patients who engaged in less exercise and physical activity had a higher risk of weight gain. Patients who underwent chemotherapy experienced a more significant decrease in exercise time (3.6 hours per week) than those who underwent surgery (1.6 hours per week). Furthermore, a study showed that all patients who underwent chemotherapy experienced amenorrhea; therefore, changes in hormones and menopause could impact metabolism, affecting body

composition and the waist-to-hip ratio. This can result in increased estrogen and insulin levels (30).

375 Oncological rehabilitation (OR) and mindfulness stimulate specific neurovascular terminals that activate ATP, improve bloodstream flow, and stimulate the 376 parasympathetic nervous system (PNS), thereby generating serotonin and 377 endorphins, relaxing muscles, improving digestion, and reducing insomnia. It also 378 prevents sarcopenia and stimulates immunoglobulins and the osteomioarticular 379 system (OMAS). Mindfulness provides a profound knowledge of the mind and its 380 discriminative processes, allowing free radicals to be dosed. Through extensive 381 382 practice, the patient learns how to regulate their attention and manages to focus on the present, which enhances the experience itself and the exercises at hand (31). 383

Psychological treatments for patients with BC indicated that cognitive behavioral and psycho-educational therapies have a significant positive impact. These therapies improved QoL, reduced anxiety and depression, and improved mood. The study found that treatment lasting between six and twelve weeks achieved better psychological results than shorter or longer interventions (32). Relaxation techniques are commonly used in mindfulness programs and psychological interventions to alleviate symptoms of depression, anxiety, stress, and fear of recurrence. Survivors of BC have reported improved sleep quality after practicing these techniques. (33). Cognitive-behavioral approaches have successfully overcome fatigue and improved sleep quality. (34). A randomized trial conducted by Rogers et al. revealed that physical activity positively impacted overall sleep quality compared to usual care in BC patients. (35).

Patients with BC have benefitted from virtual psychological interventions. One study 396 called the Web-Based Stress Management for Newly Diagnosed Patients with 397 398 Cancer (STREAM) developed an online stress management program that significantly improved the QoL for patients in the intervention group (73.2%) 399 compared to the control group (59%). The Hospital Anxiety and Depression scale 400 (HADS) score decreased, mainly due to reduced levels of distress (20). Another 401 402 study used a web-based psychological intervention called Web-Based Self-Management for Psychological Adjustment After Primary Breast Cancer (BREATH). 403 which resulted in lower levels of distress (84%) and clinical deterioration (16%) for 404 405 the intervention group (36).

#### Conclusion

384 385

386

387 388

389

390

391

392

393 394

395

406

Although there have been several studies on interventions for breast cancer patients, such as those related to nutrition, physical activity, mindfulness, or psychological support, these interventions have typically been conducted separately and focused

- 410 primarily on survivors. This highlights the necessity for multidisciplinary
- interventions, as proposed in this study.

# 412 Acknowledgments

- The authors thank the CAAI (Centro de Apoyo para la Atención Integral) of the
- 414 Instituto Nacional de Cancerología for the facilities and spaces for the
- implementation of workshops for the described intervention.

#### Contributors

416

- 417 Cruz-Ramos: protocol design, principal researcher, and draft preparation. Fajardo-
- 418 Espinoza: Protocol design, draft preparation, nutritional intervention design, and
- 419 implementation. Martinez-Palacios: Draft preparation and hybrid educational
- 420 intervention design. Pérez-Camargo: Nutritonal intervention design and
- 421 implementation. Cedillo-Compeán: Oncological rehabilitation intervention design
- and implementation. Rodríguez-Fonseca: Mindfulness specialist, hybrid educational
- intervention design and implementation. Blandón-Hernández and Labra-Alvarado:
- Psychological and Mindfulness Intervention Implementation. Gálvez-Hernández and
- Bejarano-Colina: Psychological intervention design and implementation. Villarreal-
- 426 Garza: Reviewer and protocol design. Cabrera-Nieto, Barranco-Cortés, González-
- Pérez, Madariaga-Cobos: Nutritional intervention implementation. Bargalló-Rocha,
- 428 Matus-Santos, Espinosa-Fernández and Cabrera-Galeana oncological follow-up
- 429 protocol and patient reference to the program. Mohar-Betancourt: Reviewer and
- 430 protocol design.

#### 431 Conflict of interest

- The authors declare no conflicts of interest.
- 433 Patient consent for publication. Not required

#### 434 Ethics approval

- The authors declare that this study was conducted according to the Declaration of
- 436 Helsinki, and all procedures were performed with adequate understanding and
- written consent from the individuals. The study protocol was approved by the Ethics
- 438 Committee of Instituto Nacional de Cancerología (023-005-OMI, CEI-025022).

# Funding

- None. At the time of publication, the project had not received any specific grant from
- public, commercial, or not-for-profit funding agencies or laboratories.

# Data availability statement.

443 Study results are not available yet.

444

456

- 1. Amadou A, Torres-Mejía G, Hainaut P, Romieu I. Breast cancer in Latin America: global burden, patterns, and risk factors.
- 2. Bessonneau V, Rudel RA. Mapping the human exposome to uncover the causes of breast cancer. Int J Environ Res Public Health. 2020 Jan 1;17(1).
- 3. Fang M, Hu L, Chen D, Guo Y, Liu J, Lan C, et al. Exposome in human health: Utopia or wonderland? Vol. 2, The Innovation. Cell Press; 2021.
- 4. Daiber A, Kröller-Schön S, Frenis K, Oelze M, Kalinovic S, Vujacic-Mirski K, et al. Environmental noise induces the release of stress hormones and inflammatory signaling molecules leading to oxidative stress and vascular dysfunction—Signatures of the internal exposome. Vol. 45, BioFactors. Blackwell Publishing Inc.; 2019. p. 495–506.
  - 5. Kalita-de Croft P, Sharma S, Sobrevia L, Salomon C. Extracellular vesicle interactions with the external and internal exposome in mediating carcinogenesis. Vol. 87, Molecular Aspects of Medicine. Elsevier Ltd; 2022.
- 6. Reynoso Noverón N, Villarreal Garza C, Soto Pérez de Celis E, Arce Salinas C, Matus Santos J, Ramírez Ugalde MT, et al. Clinical and Epidemiological Profile of Breast Cancer in Mexico: Results of the Seguro Popular. 2017.
- 7. Shaikh H, Bradhurst P, Ma LX, Tan SY, Egger SJ, Vardy JL. Body weight management in overweight and obese breast cancer survivors. Vol. 2020, Cochrane Database of Systematic Reviews. John Wiley and Sons Ltd; 2020.
- 8. Villarreal-Garza C, Platas A, Miaja M, Mesa-Chavez F, Garcia-Garcia M, Fonseca A, et al. Patients' satisfaction with a supportive care program for young breast cancer patients in Mexico: Joven & Fuerte supports patients' needs and eases their illness process. Supportive Care in Cancer. 2020 Oct 1;28(10):4943–51.
- 9. Bustamante-Marin XM, Merlino JL, Devericks E, Carson MS, Hursting SD, Stewart DA. Mechanistic Targets and Nutritionally Relevant Intervention

- Strategies to Break Obesity–Breast Cancer Links. Vol. 12, Frontiers in Endocrinology. Frontiers Media S.A.; 2021.
- 476 10. Ee C, Cave A, Vaddiparthi V, Naidoo D, Boyages J. Factors associated 477 with weight gain after breast cancer: Results from a community-based survey 478 of Australian women. Breast. 2023 Jun 1;69:491–8.
- 11. Nyrop KA, Deal AM, Shachar SS, Park J, Choi SK, Lee JT, et al. Weight trajectories in women receiving systemic adjuvant therapy for breast cancer. Breast Cancer Res Treat. 2020 Feb 1;179(3):709–20.
- 482 12. Perry S, Kowalski TL, Chang CH. Quality of life assessment in women 483 with breast cancer: Benefits, acceptability and utilization. Vol. 5, Health and 484 Quality of Life Outcomes. 2007.
- 485 13. Villarreal-Garza C, Águila C, Platas A, Lara-Guerra H. Cáncer de 486 mama en mujeres jóvenes en México: necesidades y retos clínicos. Revista 487 de Investigación Clínica. 2014;66(6):547–88.
- 488 14. Campbell-Enns H, Woodgate R. The psychosocial experiences of 489 women with breast cancer across the lifespan: a systematic review protocol. 490 JBI Database System Rev Implement Rep. 2015 Jan 1;13(1):112–21.
- 491 15. Montagnese C, Porciello G, Vitale S, Palumbo E, Crispo A, Grimaldi M, et al. Quality of life in women diagnosed with breast cancer after a 12-month treatment of lifestyle modifications. Nutrients. 2021 Jan 1;13(1):1–15.
- 16. Ruiz-Vozmediano J, Löhnchen S, Jurado L, Recio R, Rodríguez-Carrillo A, López M, et al. Influence of a Multidisciplinary Program of Diet, Exercise, and Mindfulness on the Quality of Life of Stage IIA-IIB Breast Cancer Survivors. Integr Cancer Ther. 2020;19.

498

499

500

- 17. Richards J, Arensberg MB, Thomas S, Kerr KW, Hegazi R, Bastasch M. Impact of early incorporation of nutrition interventions as a component of cancer therapy in adults: A review. Vol. 12, Nutrients. MDPI AG; 2020. p. 1–19.
- 502 18. Dieli-Conwright CM, Wong L, Waliany S, Bernstein L, Salehian B, 503 Mortimer JE. An observational study to examine changes in metabolic 504 syndrome components in patients with breast cancer receiving neoadjuvant or 505 adjuvant chemotherapy. Cancer. 2016 Sep 1:122(17):2646–53.

- 506 19. Snetselaar LG, de Jesus JM, DeSilva DM, Stoody EE. Dietary
- Guidelines for Americans, 2020-2025: Understanding the Scientific Process,
- Guidelines, and Key Recommendations. Nutr Today. 2021 Nov-
- 509 Dec;56(6):287-295.
- 510 20. Urech C, Grossert A, Alder J, Scherer S, Handschin B, Kasenda B, et
- al. Web-Based Stress Management for Newly Diagnosed Patients With
- 512 Cancer (STREAM): A Randomized, Wait-List Controlled Intervention Study. J
- 513 Clin Oncol [Internet]. 2018;36:780–8. Available from:
- 514 https://doi.org/10.1200/JCO.2017.
- 515 21. Fowler S. Diabetes Prevention Program (V8) [Dataset]. NIDDK Central
- 516 Repository. 2023;
- 517 22. Hauner D, Rack B, Friedl T, Hepp P, Janni W, Hauner H. Rationale
- and description of a lifestyle intervention programme to achieve moderate
- weight loss in women with non-metastatic breast cancer: The lifestyle
- intervention part of the SUCCESS C Study. BMJ Nutr Prev Health. 2020 Dec
- 521 1;3(2):213–9.
- 522 23. Di Meglio A, Martin E, Crane TE, Charles C, Barbier A, Raynard B, et
- al. A phase III randomized trial of weight loss to reduce cancer-related fatigue
- among overweight and obese breast cancer patients: MEDEA Study design.
- 525 Trials. 2022 Dec 1;23(1).
- 526 24. Febvey-Combes O, Jobard E, Rossary A, Pialoux V, Foucaut AM,
- Morelle M, et al. Effects of an Exercise and Nutritional Intervention on
- 528 Circulating Biomarkers and Metabolomic Profiling During Adjuvant Treatment
- for Localized Breast Cancer: Results From the PASAPAS Feasibility
- Randomized Controlled Trial. Integr Cancer Ther. 2021;20.
- 1. Amadou A, Torres-Mejía G, Hainaut P, Romieu I. Breast cancer in
- Latin America: global burden, patterns, and risk factors.
- 533 2. Bessonneau V, Rudel RA. Mapping the human exposome to uncover
- the causes of breast cancer. Int J Environ Res Public Health. 2020 Jan 1;17(1).
- 535 3. Fang M, Hu L, Chen D, Guo Y, Liu J, Lan C, et al. Exposome in human
- health: Utopia or wonderland? Vol. 2, The Innovation. Cell Press; 2021.
- 537 4. Daiber A, Kröller-Schön S, Frenis K, Oelze M, Kalinovic S, Vujacic-
- 538 Mirski K, et al. Environmental noise induces the release of stress hormones
- and inflammatory signaling molecules leading to oxidative stress and vascular

- 540 dysfunction—Signatures of the internal exposome. Vol. 45, BioFactors. 541 Blackwell Publishing Inc.; 2019. p. 495–506.
- 5. Kalita-de Croft P, Sharma S, Sobrevia L, Salomon C. Extracellular vesicle interactions with the external and internal exposome in mediating carcinogenesis. Vol. 87, Molecular Aspects of Medicine. Elsevier Ltd; 2022.
- 545 6. Reynoso Noverón N, Villarreal Garza C, Soto Pérez de Celis E, Arce 546 Salinas C, Matus Santos J, Ramírez Ugalde MT, et al. Clinical and 547 Epidemiological Profile of Breast Cancer in Mexico: Results of the Seguro 548 Popular. 2017.
- 7. Shaikh H, Bradhurst P, Ma LX, Tan SY, Egger SJ, Vardy JL. Body weight management in overweight and obese breast cancer survivors. Vol. 2020, Cochrane Database of Systematic Reviews. John Wiley and Sons Ltd; 2020.
- 553 8. Villarreal-Garza C, Platas A, Miaja M, Mesa-Chavez F, Garcia-Garcia M, Fonseca A, et al. Patients' satisfaction with a supportive care program for young breast cancer patients in Mexico: Joven & Fuerte supports patients' needs and eases their illness process. Supportive Care in Cancer. 2020 Oct 1;28(10):4943–51.
- 558 9. Bustamante-Marin XM, Merlino JL, Devericks E, Carson MS, Hursting 559 SD, Stewart DA. Mechanistic Targets and Nutritionally Relevant Intervention 560 Strategies to Break Obesity–Breast Cancer Links. Vol. 12, Frontiers in 561 Endocrinology. Frontiers Media S.A.; 2021.
- 562 10. Ee C, Cave A, Vaddiparthi V, Naidoo D, Boyages J. Factors associated 563 with weight gain after breast cancer: Results from a community-based survey 564 of Australian women. Breast. 2023 Jun 1;69:491–8.
- 565 11. Nyrop KA, Deal AM, Shachar SS, Park J, Choi SK, Lee JT, et al. Weight trajectories in women receiving systemic adjuvant therapy for breast cancer. Breast Cancer Res Treat. 2020 Feb 1;179(3):709–20.
- 568 12. Perry S, Kowalski TL, Chang CH. Quality of life assessment in women with breast cancer: Benefits, acceptability and utilization. Vol. 5, Health and Quality of Life Outcomes. 2007.
- 571 13. Villarreal-Garza C, Águila C, Platas A, Lara-Guerra H. Cáncer de 572 mama en mujeres jóvenes en México: necesidades y retos clínicos. Revista 573 de Investigación Clínica. 2014;66(6):547–88.

- 574 14. Campbell-Enns H, Woodgate R. The psychosocial experiences of women with breast cancer across the lifespan: a systematic review protocol.
  576 JBI Database System Rev Implement Rep. 2015 Jan 1;13(1):112–21.
- 577 15. Montagnese C, Porciello G, Vitale S, Palumbo E, Crispo A, Grimaldi M, et al. Quality of life in women diagnosed with breast cancer after a 12-month treatment of lifestyle modifications. Nutrients. 2021 Jan 1;13(1):1–15.
- 16. Ruiz-Vozmediano J, Löhnchen S, Jurado L, Recio R, Rodríguez-Carrillo A, López M, et al. Influence of a Multidisciplinary Program of Diet, Exercise, and Mindfulness on the Quality of Life of Stage IIA-IIB Breast Cancer Survivors. Integr Cancer Ther. 2020;19.
- 17. Richards J, Arensberg MB, Thomas S, Kerr KW, Hegazi R, Bastasch M. Impact of early incorporation of nutrition interventions as a component of cancer therapy in adults: A review. Vol. 12, Nutrients. MDPI AG; 2020. p. 1–19.
- 588 18. Dieli-Conwright CM, Wong L, Waliany S, Bernstein L, Salehian B,
  589 Mortimer JE. An observational study to examine changes in metabolic
  590 syndrome components in patients with breast cancer receiving neoadjuvant or
  591 adjuvant chemotherapy. Cancer. 2016 Sep 1;122(17):2646–53.
- 19. U.S. Department of Agriculture. https://www.myplate.gov/. My Plate.
- 20. Urech C, Grossert A, Alder J, Scherer S, Handschin B, Kasenda B, et 593 al. Web-Based Stress Management for Newly Diagnosed Patients With 594 Cancer (STREAM): A Randomized, Wait-List Controlled Intervention Study. J 595 Clin Oncol [Internet]. 2018;36:780–8. Available from: 596 https://doi.org/10.1200/JCO.2017. 597
- 598 21. Fowler S. Diabetes Prevention Program (V8) [Dataset]. NIDDK Central Repository. 2023;
- Hauner D, Rack B, Friedl T, Hepp P, Janni W, Hauner H. Rationale and description of a lifestyle intervention programme to achieve moderate weight loss in women with non-metastatic breast cancer: The lifestyle intervention part of the SUCCESS C Study. BMJ Nutr Prev Health. 2020 Dec 1;3(2):213–9.
- Di Meglio A, Martin E, Crane TE, Charles C, Barbier A, Raynard B, et al. A phase III randomized trial of weight loss to reduce cancer-related fatigue

- among overweight and obese breast cancer patients: MEDEA Study design.
- 608 Trials. 2022 Dec 1;23(1).
- 609 24. Febvey-Combes O, Jobard E, Rossary A, Pialoux V, Foucaut AM,
- Morelle M, et al. Effects of an Exercise and Nutritional Intervention on
- 611 Circulating Biomarkers and Metabolomic Profiling During Adjuvant Treatment
- for Localized Breast Cancer: Results From the PASAPAS Feasibility
- Randomized Controlled Trial. Integr Cancer Ther. 2021;20.
- Batsis JA, McClure AC, Weintraub AB, Sette D, Rotenberg S, Stevens
- 615 CJ, et al. Barriers and facilitators in implementing a pilot, pragmatic,
- telemedicine-delivered healthy lifestyle program for obesity management in a
- rural, academic obesity clinic. Implement Sci Commun. 2020 Dec 1;1(1).
- 618 26. King DK, Shoup JA, Raebel MA, Anderson CB, Wagner NM, Ritzwoller
- DP, et al. Planning for Implementation Success Using RE-AIM and CFIR
- Frameworks: A Qualitative Study. Front Public Health. 2020 Mar 3;8.
- De Cicco P, Catani MV, Gasperi V, Sibilano M, Quaglietta M, Savini I.
- Nutrition and breast cancer: A literature review on prevention, treatment and
- recurrence. Vol. 11, Nutrients. MDPI AG; 2019.
- 624 28. Hoy MK, Winters BL, Chlebowski RT, Papoutsakis C, Shapiro A, Lubin
- MP, et al. Implementing a Low-Fat Eating Plan in the Women's Intervention
- 626 Nutrition Study. J Am Diet Assoc. 2009 Apr;109(4):688–96.
- 29. Demark-Wahnefried W. Reduced rates of metabolism and decreased
- 628 physical activity in breast cancer patients receiving adjuvant chemotherapy 1 3
- 629 [Internet]. Vol. 65. 1997. Available from:
- https://academic.oup.com/ajcn/article-abstract/65/5/1495/4655500
- 631 30. Makari-Judson G, Braun B, Joseph Jerry D, Mertens WC. Weight gain
- following breast cancer diagnosis: Implication and proposed mechanisms. Vol.
- 5, World Journal of Clinical Oncology. Baishideng Publishing Group Co.,
- 634 Limited; 2014. p. 272–82.
- 635 31. Kabat-Zinn J. Mindfulness-based interventions in context: Past,
- present, and future. Vol. 10, Clinical Psychology: Science and Practice. 2003.
- 637 p. 144–56.
- 638 32. Guarino A, Polini C, Forte G, Favieri F, Boncompagni I, Casagrande
- M. The effectiveness of psychological treatments in women with breast cancer:

- A systematic review and meta-analysis. Vol. 9, Journal of Clinical Medicine. MDPI; 2020.
- 33. Lengacher CA, Reich RR, Paterson CL, Shelton M, Shivers S, Ramesar S, et al. A Large Randomized Trial: Effects of Mindfulness-Based Stress Reduction (MBSR) for Breast Cancer (BC) Survivors on Salivary Cortisol and IL-6. Biol Res Nurs. 2019 Jan 1;21(1):39–49.
- 34. Widiasih R, Ermiati, Jayanti TN, Rais Y. Psychosocial Interventions for
   Improving the Quality of Life in Breast Cancer Survivors: A Literature Review.
   In: IOP Conference Series: Earth and Environmental Science. Institute of
   Physics Publishing; 2019.
- 650 35. Rogers LQ, Courneya KS, Oster RA, Anton PM, Robbs RS, Forero A, 651 et al. Physical activity and sleep quality in breast cancer survivors: A 652 randomized trial. Med Sci Sports Exerc. 2017 Oct 1;49(10):2009–15.
- 36. Van Den Berg SW, Gielissen MFM, Custers JAE, Van Der Graaf WTA,
  Ottevanger PB, Prins JB. BREATH: Web-based self-management for
  psychological adjustment after primary breast cancer-results of a multicenter
  randomized controlled trial. Journal of Clinical Oncology. 2015 Sep
  1;33(25):2763–71.